CLINICAL TRIAL: NCT07405905
Title: MINI IMPLANTS PLACED AT INFRAZYGOMATIC CREST VERSUS INTERRADICULAR SITES A RANDOMIZED CLINICAL TRIAL.
Brief Title: EVALUATION OF TREATMENT CHANGES IN CLASS II DIVISION 1 MALOCCLUSION DURING EN MASSE RETRACTION OF UPPER ANTERIOR TEETH USING MINI IMPLANTS PLACED AT INFRAZYGOMATIC CREST AND INTERRADICULAR SITES A RANDOMIZED CLINICAL TRIAL.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SONAL NAYAN
Record Dates: First submitted 2026-01-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: CLASS II DIVISION 1 MALOCCLUSION
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retraction of anterior teeth using mini implants placed at infrazygomatic crest. (Experimental): bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at infrazygomatic crest
  Interventions: Procedure: retraction of anterior teeth using mini implants placed at infrazygomatic crest.
- Retraction of anterior teeth using mini implants placed at interradicular sites. (Experimental): bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at interradicular sites.
  Interventions: Procedure: retraction of anterior teeth using mini implants placed at interradicular sites.

INTERVENTIONS:
Procedure: retraction of anterior teeth using mini implants placed at infrazygomatic crest. — undergo bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at infrazygomatic crest.
  Arms: Retraction of anterior teeth using mini implants placed at infrazygomatic crest.
Procedure: retraction of anterior teeth using mini implants placed at interradicular sites. — bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at interradicular sites.
  Arms: Retraction of anterior teeth using mini implants placed at interradicular sites.

SUMMARY:
Rationale: Class II Division 1 malocclusion is characterized by upper anterior teeth protrusion resulting in upper lip protrusion and convex facial profile, which are considered esthetically unfavorable. Treatment of class II malocclusion due to maxillary protrusion can be done with bilateral maxillary first premolar extraction followed by en-masse retraction of upper anterior teeth using mini-implants placed at infrazygomatic or interradicular sites.

Aims and Objectives: To evaluate the treatment changes achieved in class II division 1 malocclusion during en- masse retraction of upper anterior teeth using mini-implants placed at infrazygomatic crest versus interradicular sites.

To compare patients' and orthodontist's perceptions of treatment being done in both the groups.

Method of study: Treatment will be initiated by bilateral maxillary 1st premolar extraction followed by bonding 0.022" slot MBT preadjusted edgewise appliance. Maxillary arch will be stabilized with the help of 0.019"×0.025" stainless steel wire and then randomized allocation of the patients into 2 groups-G1 and G2 will be done. G1 will receive infrazygomatic crest mini-implants bilaterally and G2 will receive bilateral interradicular mini-implants. Hooks will be soldered on archwire used for stabilizing dentition. Ni-Ti closed coil spring will be used to apply force.

DETAILED DESCRIPTION:
The present study is a randomized clinical trial , non-pharmacological, double blind, to evaluate the treatment changes achieved in class II division 1 malocclusion during en-masse retraction of upper anterior teeth using mini-implants placed at infrazygomatic crest versus interradicular sites. The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopaedics, in conjunction with the Department of Oral and Maxillofacial Surgery, P.G.I.D.S., Pt. B.D.Sharma University of Health Sciences, Rohtak. The study will be carried out after the institutional approval obtained from the ethical committee.

Inclusion criteria:- Non growing patients with bilateral Class II molar relationship at pre-treatment, all permanent teeth upto the second molars should be present, no or minor crowding in the maxillary arch, horizontal to average growth pattern.

Exclusion Criteria:- Subjects with a history of fixed orthodontic treatment, crossbite, vertical growth pattern, any systemic disease affecting bone and general growth, poor oral hygiene, cleft patients, patients who fail to follow up or undergo complete treatment.

INFORMED CONSENT OF THE PATIENT AND AGREEMENT TO BE RANDOMIZED A valid, written informed consent of the patient or parent/ guardian and an agreement to be randomized will be obtained from the patient before registering the patient in this clinical study. Patient will be informed about all the theoretical risks and benefits of the intervention under test . The patient will be given 72 hours to discuss the study with his/her family and take the decision regarding participation in the study.

RANDOMIZATION & ALLOCATION CONCEALMENT Randomization will be done by a person not involved in the trial using computer generated randomization list. The study subjects will be blinded regarding intervention group.

INTERVENTION AND DESIGN OF STUDY The main intervention in this prospective clinical study is the bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini-implants placed at infrazygomatic crest in group 1 (G1) and mini-implants placed at interradicular sites in group 2 (G2). The study consists of 2 groups with equal allocation of subjects in each group:- Group 1 (G1):- This group will undergo bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at infrazygomatic crest.

Group 2 (G2):- This group will undergo bilateral extraction of maxillary first premolars before initial leveling and alignment followed by retraction of anterior teeth using mini implants placed at interradicular sites.

DATA COLLECTION The investigator will record the patient's name, address and contact number will be taken. Cephalometric radiographs will be recorded before placement of mini-implants and after 6 months of application of NiTi closed coil springs. These cephalometric radiographs will be analyzed and the relevant values will be entered in a predesigned format.

Patients will be asked to fill a questionnaire in which they will be asked about problems they might have while eating, talking ,laughing, yawning swallowing ,drinking ,brushing and also the pain experienced in tooth ,jaws, muscles, headache, swelling ,soft tissue ulceration ,restricted mouth opening ,and level of satisfaction .These questionnaires will be completed on the evening after force application and at 7 days ,14 days ,1 month and 6 months. .

In addition orthodontist's perceptions will be assessed during handling complexity of mini implant in both the positions on same day,1 month, 3 months and 6 months following orthodontic force application.

STATISTICAL ANALYSIS The data entered will be processed by standard statistical analysis. Results will be presented in the form of tables and graphs.

The data will be subjected to descriptive analysis for mean, standard deviation for quantitative and proportion for qualitative variables. Shapiro Wilk test will be used to check the normality of distribution.

Independent T test (normal distribution) and Mann Whitney U test (Non-normal distribution ) will be used to compare means between two groups at pre-retraction stage. Dependent T test (normal distribution) or Wilcoxon Signed Ranks(Non-normal distribution) test will be used to compare changes within groups. Independent T test and Mann Whitney U tests will be used to compare change between two groups i.e. Group 1 (Infrazygomatic mini-implant) and Group 2 (Interradicular mini-implant). In all the analysis, the level of significance will be set a 5 percent.

Patient pain perception and orthodontist perception regarding treatment has been evaluated using chi square test.

ELIGIBILITY:
Inclusion Criteria:

1. Non growing patients
2. Bilateral Class II molar relationship at pre-treatment.
3. All permanent teeth upto the second molars should be present.
4. No or minor crowding in the maxillary arch.
5. Horizontal to average growth pattern.

Exclusion Criteria:

1. Subjects with a history of fixed orthodontic treatment.
2. Crossbite
3. Vertical growth pattern
4. Any systemic disease affecting bone and general growth
5. Poor oral hygiene
6. Cleft patients
7. Patients who fail to follow up or undergo complete treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
skeletal and dental cephalometric variables | 15 months
  Comparison of pretreatment and post 6 month evaluation of skeletal and dental cephalometric variables between the two groups Skeletal cephalometric variables
  1. SNA: SN to NA angle
  2. A-NPerp: linear distance from A-point to nasion-perpendicular(a line perpendicular to Frankfort plane, through nasion)
  3. SNB: SN to NB angle
  4. SND: SN to ND angle
  5. LAFH (lower anterior face height): distance from anterior nasal spine to menton.
  Dental cephalometric variables
  1. Mx1.NA: maxillary incisor long axis to NA angle
  2. Mx1-NA: distance between the maxillary central incisor edge and the NA line
  3. Mx1-VRL: distance from the maxillary central incisor edge to VRL (vertical reference line passing through sella and perpendicular to horizontal line constructed by reducing 7° from SN line)
  4. Mx6-VRL: distance from maxillary first molar mesial cusp to VRL
  5. Md1.NB: mandibular incisor long axis to NB angle
  6. Md1-NB: distance between the mandibular central incisor edge and the NB line.

SECONDARY OUTCOMES:
soft tissue variables between the two groups | 15 months
  Comparison of pretreatment and post 6 month evaluation of soft tissue variables between the two groups
  1. LL-E plane: distance from the lower lip to the esthetic plane of Ricketts (line from Pg= to Pr)
  2. UL-E plane: distance from the upper lip to the esthetic plane of Ricketts
  3. UL-S line: distance from the upper lip to Steiner's S line (line from Pg= to Cl)
  4. LL-S line: distance from the lower lip to Steiner's S line
  5. UL-SnPg: distance from the upper lip to the subnasale-soft-tissue pogonion plane (line from Sn to Pg)
  6. LL-SnPg: distance from the lower lip to the subnasale-soft-tissue pogonion plane
  7. H.NB: H line (tangent to Pg= and UL) to NB line angle
  8. H-Pr: distance between H line and the most anterior point on the nose
  9. Nasolabial angle: Cl.Sn.UL angle

OTHER OUTCOMES:
patient attitude and pain perception | 15 months
  Questionnaire for evaluating patient attitude and pain perception for orthodontic treatment
  1. Did your doctor in terms of pain/discomfort and its impact explain you properly about the appliance on daily activity? Yes No
  2. Did you feel embarrassment/discomfort in front of others while talking?
     (a) Not at all (b) a little (c) a lot (d) does not worry me
  3. Did you feel embarrassment/discomfort in front of other while eating?
     (a) Not at all (b) a little (c) a lot (d) does not worry me
  4. Did you get any soft tissue lacerations?
     (a) Receiving of the appliance (b) Using the appliance (c) Breakage of appliance (d) None of the above
  5. Did you ask the doctor to remove the appliance because you felt it is too hard to have it in your mouth for the long time? Yes No
orthodontic perception | 15 months
  Questionare for orthodontic perception during treatment
  1. Handling complexity of mini-implant attachment
     a)very easy b)easy c)somewhat easy d)difficult e)very difficult
  2. Mobility
     a)no b)mild c)moderate that treatment discontinued for sometime d)severe that treatment stopped
  3. soft tissue ulcer
  4. fracture
  5. undesirable position
  6. infection

CONTACTS AND LOCATIONS:
Overall Officials: Sonal chowdhary, MDS, Study Director — Post Graduate Institute of Dental Sciences, Rohtak, Haryana 124001 Recruiting
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana 124001, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol